CLINICAL TRIAL: NCT03201445
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Testicular Safety of Filgotinib in Adult Males With Moderately to Severely Active Inflammatory Bowel Disease
Brief Title: Study to Evaluate the Testicular Safety of Filgotinib in Adult Males With Moderately to Severely Active Inflammatory Bowel Disease
Acronym: MANTA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early Termination for Reasons other than Safety
Sponsor: Galapagos NV (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-418-4279; 2017-000402-38 (EudraCT Number)
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — GLPG0634; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Filgotinib (Experimental): Participants received filgotinib up to Week 13 in the DB phase (Part A). At Week 13, participants who were IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB treatment up to Week 26 (Part B). Participants who were IBD non-responders at Week 13 or had disease worsening after Week 13 and prior to Week 26, and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib for up to Week 13. At Week 26/OL Week 13, participants who were IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet a prespecified decrease threshold, continued receiving the same study drug they were responding to as part of the LTE for up to 195 weeks. Participants who met pre-specified sperm decrease threshold(s) at any postbaseline visit discontinued study drug and switched to a standard of care (SOC) regimen selected by the investigator and entered the MP for up to 52 weeks.
  Interventions: Drug: Filgotinib; Drug: Standard of Care
- Placebo (Placebo Comparator): Participants received placebo (matched to filgotinib) up to Week 13 in the DB phase (Part A). At Week 13, participants who were IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB treatment up to Week 26 (Part B). Participants who were IBD non-responders at Week 13 or had disease worsening after Week 13 and prior to Week 26, and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib for up to Week 13. At Week 26/OL Week 13, participants who were IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet a prespecified decrease threshold, continued receiving the same study drug they were responding to as part of the LTE for up to 195 weeks. Participants who met pre-specified sperm decrease threshold(s) at any postbaseline visit discontinued study drug and switched to SOC regimen selected by the investigator and entered the MP for up to 52 weeks.
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Filgotinib — 200 mg tablet administered orally once daily
  Arms: Filgotinib
Drug: Placebo — Placebo to match filgotinib tablet administered orally once daily
  Arms: Placebo
Drug: Standard of Care — Locally approved treatment, accepted by medical experts as a proper treatment for IBD conditions, prescribed according to best clinical practice, with no known testicular toxicity.

SUMMARY:
The primary objective of this study is to evaluate the testicular safety of filgotinib in adult males with moderately to severely active inflammatory bowel disease (IBD).

Results of this study may be pooled with the results of a separate study being conducted in participants with rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or non-radiographic axial spondyloarthritis (Protocol GLPG0634-CL-227; NCT03926195) with the same objective. The total planned number of participants in both studies combined will be up to approximately 250 participants.

DETAILED DESCRIPTION:
There are 5 parts to the study: 1) Part A: Double-Blind Phase (DB Phase; Day 1 through Week 13); 2) Part B: DB Phase (after Week 13 through Week 26); 3) Open-label (OL) Filgotinib Phase (after Week 13 study visit for up to 13 weeks); 4) Monitoring Phase (MP; up to 52 weeks); and 5) Long-term Extension (LTE) Phase (after Week 26 or end of OL Filgotinib Phase for up to 195 weeks).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of ulcerative colitis (UC) or Crohn's Disease (CD) of at least 4 months. Endoscopic and histopathologic documentation of UC or CD.
* Have moderately to severely active UC or CD

Key Exclusion Criteria:

* Previously or currently documented problems with male reproductive health
* Current use of sulfasalazine or its use within the 26 weeks leading up to Screening; sulfasalazine is not permitted at any point during the study
* Current use of corticosteroids at a dosage of > 20 mg/day of prednisone or equivalent at randomization
* Indeterminate colitis, ischemic colitis, fulminant colitis, isolated ulcerative proctitis, or toxic mega colon
* Active tuberculosis (TB) or untreated latent tuberculosis
* Use of concomitant prohibited medications as outlined by protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2023-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (56):
- United States (10):
  - Naval Medical Center San Diego, San Diego, California
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - One Health Research Clinic, Inc, Norcross, Georgia
  - Delta Research Partners, Monroe, Louisiana
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastro One, Germantown, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
- Monash Medical Centre, Clayton, Victoria, Australia
- AKH Wien - Universitatsklinik fur Innere Medizin III, Vienna, Austria
- Medizinische Hochschule Hannover, Hanover, Germany
- India (23):
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Seth GS medical college and KEM hospital, Pārel, Mumbai
  - Kaizen Hospital, Ahmedabad
  - SP Medical college & AG Hospitals, Bīkaner
  - Maharaja Agrasen Hospital, Dehli
  - Nizam's Institute of Medical Sciences, Hyderabad
  - SR Kalla Memorial Gastro and General Hospital, Jaipur
  - SMS Medical College and Hospital, Jaipur
  - Om Sai Onco Surgery Center, Kolhāpur
  - Institute of Post Graduate Medical Education and Research (IPGMER), Kolkata
  - Radha Krishna Critical Care & General Hospital, Kota
  - Dayanand Medical College & Hospital, Ludhiana
  - Rahate Surgical Hospital, Nagpur
  - Crescent Hospital and Heart Centre, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Batra Hospital and Medical Research Center, New Delhi
  - Shri Griraj Multispeciality Hospital, Rajkot
  - Gandhi Hospital, Secunderabad
  - Institute of Gastroenterology & Liver Disease, Sunshine Hospitals, Secunderabad
  - BAPS Pramukh Swami Hospital, Surat
  - Sterling Hospital, Vadodara
  - Samvedna Hospital, Varanasi
- Wellington Hospital, Newtown, New Zealand
- Poland (5):
  - Osrodek Badan Klinicznych Cinsante S.C Ewa Galczak-Nowak, Bydgoszcz
  - Krakowskie Centrum Medyczne, Krakow
  - Santa Familia, Centrum Badan Profilaktyki i Leczenia, Lodz
  - Endoskopia Sp.z o.o, Sopot
  - Bodyclinic Alicja Pasnik, Warsaw
- S.C. Policlinica Dr. Citu S.R.L - Gastroenterologie, Timișoara, Romania
- Russia (4):
  - Olla-Med, Llc, Moscow
  - State Budgetary Healthcare Institution, Pensa Regional Clinical Hospital n.a N.N Burdenko, Penza
  - State Budgetary Educational Institution of Higher Professional Education "Rostov State Medical University" of the Ministry of Health of Russian Fedn., Rostov-on-Don
  - Saint Petersburg State Budgetary Healthcare Institution "City Hospital # 26", Saint Petersburg
- Ukraine (8):
  - Municipal Health Care Institution "Regional Hospital of War Veterans", Therapeutic Department No. 1, Kharkiv
  - Kyiv City Clinical Hospital #18, Proctology Department, Kiev
  - Vinnytsia Regional Clinical Hospital of War Veterans, Therapeutics Department No. 2, Vinnitsa
  - Vinnytsia Regional Clinical Hospital named after M.I. Pirogov, Gastroenterology Department, Vinnitsya
  - Medical Center LLC "Health Clinic", Medical Clinical Investigational Center, Vinnitsya
  - Vinnytsia Regional Clinical Hospital of War Veterans, Therapeutics Department No.1, Vinnytsia
  - Municupal Institution "Zaporizhzhia City Multidisciplinary Clinic #9" Gastrointestinal Surgery Department,, Zaporizhzhya
  - Municipal Non-profit Enterprise "Zaporizhzhia Regional Clinical Hospital" of Zaporizhzhia Regional Council,, Zaporizhzhya
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinisch W, Hellstrom W, Dolhain RJEM, Sikka S, Westhovens R, Mehta R, Ritter T, Seidler U, Golovchenko O, Simanenkov V, Garmish O, Jeka S, Moravcova R, Rajendran V, Le Brun FO, Arterburn S, Watkins TR, Besuyen R, Vanderschueren D. Effects of filgotinib on semen parameters and sex hormones in male patients with inflammatory diseases: results from the phase 2, randomised, double-blind, placebo-controlled MANTA and MANTA-RAy studies. Ann Rheum Dis. 2023 Aug;82(8):1049-1058. doi: 10.1136/ard-2023-224017. Epub 2023 May 3. PMID 37137672
- [Derived] Hellstrom WJG, Dolhain RJEM, Ritter TE, Watkins TR, Arterburn SJ, Dekkers G, Gillen A, Tonussi C, Gilles L, Oortwijn A, Van Beneden K, de Vries DE, Sikka SC, Vanderschueren D, Reinisch W. MANTA and MANTA-RAy: Rationale and Design of Trials Evaluating Effects of Filgotinib on Semen Parameters in Patients with Inflammatory Diseases. Adv Ther. 2022 Jul;39(7):3403-3422. doi: 10.1007/s12325-022-02168-4. Epub 2022 May 25. PMID 35614292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Austria, Germany, India, New Zealand, Poland, Romania, Russian Federation, Ukraine, United Kingdom, and United States. The first participant was screened on 11 July 2017. A total of 323 participants were screened of which 139 participants were randomized into the study.
Pre-assignment Details: Study had 5 parts: Part A: Double-Blind Phase (DB Phase; Day 1 up to Week 13); Part B: DB Phase (Week 13 up to Week 26); Open-label (OL) Phase (after Week 13 study visit for up to 13 weeks); Monitoring Phase (MP; up to 52 weeks); and Long-term Extension (LTE) Phase (after Week 26 or end of OL Phase for up to 195 weeks).
Groups:
- Filgotinib: Participants received filgotinib 200 milligrams (mg) tablet, orally, once daily up to Week 13 in the DB phase (Part A). At Week 13, participants who were inflammatory bowel disease (IBD) responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B). Participants who were IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib 200 mg, tablet, orally, once daily for up to Week 13 during the OL phase. At Week 26/OL Week 13, participants who were IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet a prespecified decrease threshold, continued receiving the same study drug they were responding to (ie, blinded study drug or OL filgotinib) as part of the LTE for up to 195 weeks. Participants who met pre-specified sperm decrease threshold(s) at any postbaseline visit discontinued study drug and switched to a standard of care (SOC) regimen selected by the investigator (in accordance with the protocol) and entered the MP for up to 52 weeks.
- Placebo: Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase (Part A). At Week 13, participants who were IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B). Participants who were IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib 200 mg, tablet, orally, once daily for up to Week 13 during the OL phase. At Week 26/OL Week 13, participants who were IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet a prespecified decrease threshold, continued receiving the same study drug they were responding to (ie, blinded study drug or OL filgotinib) as part of the LTE for up to 195 weeks. Participants who met pre-specified sperm decrease threshold(s) at any postbaseline visit discontinued study drug and switched to SOC regimen selected by the investigator (in accordance with the protocol) and entered the MP for up to 52 weeks.
Period: Part A DB Phase (Through Week 13)
Arm/Group | Filgotinib | Placebo
Started | 69 | 70
Completed | 68 | 67
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Part B DB Phase (Week 13 to 26)
Arm/Group | Filgotinib | Placebo
Started | 45 (45 participants continued DB after Week 13, 1 participant switched to MP, 22 participants switched to OL) | 38 (38 participants continued DB after Week 13, 6 participants switched to MP, 23 participants switched to OL)
Completed | 42 (38 participants continued DB after Week 26, 2 participants stopped DB study drug at Week 26, 2 participants switched to MP) | 38 (34 participants continued DB after Week 26, 1 participant stopped DB study drug at Week 26, 3 participants switched to MP)
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Progressive Disease | 2 | 0
Period: OL Phase (13 Weeks)
Arm/Group | Filgotinib | Placebo
Started | 24 (2 additional participants in the Filgotinib group who were responders discontinued study drug between Weeks 13 and 26 due to disease worsening and switched to OL filgotinib, per protocol.) | 23
Completed | 22 (18 participants continued OL filgotinib in LTE, 3 participants stopped OL filgotinib in LTE, 1 participant switched to MP) | 20 (16 participants continued OL filgotinib in LTE, 2 participants stopped OL filgotinib in LTE, 2 participant switched to MP)
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Period: LTE: DB Study Drug (up to Week 195)
Arm/Group | Filgotinib | Placebo
Started (Participants who continued DB study drug after Week 26 (IBD responder and did not meet sperm decrease threshold) in the LTE.) | 38 | 34
Completed | 8 | 5
Not Completed | 30 | 29
Not completed — Adverse Event | 9 | 10
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Pre-Specified Decrease In Sperm Parameters (Switched to MP) | 6 | 7
Not completed — Study Terminated By Sponsor | 11 | 5
Period: LTE: OL Study Drug (Up to Week 195)
Arm/Group | Filgotinib | Placebo
Started (Participants who continued OL filgotinib (IBD responder and did not meet sperm decrease threshold) in the LTE.) | 18 | 16
Completed | 0 | 2
Not Completed | 18 | 14
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pre-Specified Decrease In Sperm Parameters (Switched to MP) | 5 | 3
Not completed — Progressive Disease | 2 | 0
Not completed — Study Terminated By Sponsor | 6 | 6
Period: Monitoring Phase (Up to Week 52)
Arm/Group | Filgotinib | Placebo
Started (The participants who experienced a ≥50% decrease in sperm concentration, and/or motility, and/or morphology at any time at/after 13 weeks on study drug, discontinued study drug and switched to standard of care, and started the MP.) | 15 (1 participant at Week 13 , 3 participants at Week 26/OL Week 13, and 11 participants at/after Week 39/OL Week 26 entered the MP.) | 21 (6 participants at Week 13 , 5 participants at Week 26/OL Week 13, and 10 participants at/after Week 39/OL Week 26 entered the MP.)
Completed | 14 | 19
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated By Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who took ≥ 1 dose of double-blind study drug.
Groups:
- Filgotinib: Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase (Part A). At Week 13, participants who were IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B). Participants who were IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib 200 mg, tablet, orally, once daily for up to Week 13 during the OL phase. At Week 26/OL Week 13, participants who were IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet a prespecified decrease threshold, continued receiving the same study drug they were responding to (ie, blinded study drug or OL filgotinib) as part of the LTE for up to 195 weeks. Participants who met pre-specified sperm decrease threshold(s) at any postbaseline visit discontinued study drug and switched to a SOC regimen selected by the investigator (in accordance with the protocol) and entered the MP for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Filgotinib | Placebo | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8.5) | 34 (8.4) | 35 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 69 | 70 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 68 | 68 | 136
    Ethnicity: Hispanic or Latino | 1 | 1 | 2
    Ethnicity: Not Permitted | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 2 | 0 | 2
    Race: Asian | 37 | 38 | 75
    Race: Black or African American | 1 | 0 | 1
    Race: White | 29 | 31 | 60
    Race: Not Permitted | 0 | 1 | 1
Sperm Concentration [Mean (Standard Deviation); unit: million sperm cells/milliliter (mL)] | 63.4 (34.34) | 61.8 (34.96) | 62.6 (34.53)
Total Sperm Count [Mean (Standard Deviation); unit: million sperm cells/ejaculate] | 190.6 (107.08) | 171.1 (100.74) | 180.8 (104.02)
Sperm Total Motility [Mean (Standard Deviation); unit: percentage of motile sperm] | 59.6 (11.33) | 58.6 (10.94) | 59.1 (11.11)
Ejaculate Volume [Mean (Standard Deviation); unit: mL] | 3.2 (1.20) | 3.0 (1.48) | 3.1 (1.35)
Percent Normal Sperm Morphology [Mean (Standard Deviation); unit: percentage of normal sperm] | 41 (6.4) | 41 (5.5) | 41 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 50% Decrease From Baseline in Sperm Concentration at Week 13
Description: Baseline for sperm/semen parameters was the mean of 2 evaluable semen samples at screening. The normal range for sperm concentration is ≥15 million sperm cells/mL. Percentage change = ([mean at Week 13 - baseline] / baseline) × 100; value at Week 13 was the mean of 2 evaluable samples collected at Week 13.
Time Frame: Baseline to Week 13
Population: The Semen Analysis Set included all randomized and treated (≥ 1 dose of double-blind study drug) participants who had 2 semen samples that were eligible for mean calculation at baseline and at the Week 13 analysis visit with the date of the first chronologic semen sample used for purposes of assigning analysis visit windows.
Measure: Number; unit: percentage of participants
Groups:
- Filgotinib: Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase (Part A).
- Placebo: Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase (Part A).
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 66 | 67
percentage of participants | 1.5 | 9.0
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Other; Difference in Percentage = -7.8, 95% CI 2-sided [-16.3 to 0.7] — Difference in percentage and 95% confidence interval (CI) was based on a stratified Mantel-Haenszel test

2. Secondary Outcome: Percentage of Participants With a ≥ 50% Decrease From Baseline in Sperm Concentration at Week 26
Description: IBD responder: For ulcerative colitis (UC), a participant who had a reduction of ≥2 in partial Mayo Clinic Score (pMCS) compared with baseline at specified time. For Crohn's disease (CD), a participant who had a reduction of ≥100 points in total Crohn's Disease Activity Index (CDAI) score compared with baseline at specified time. A participant with a baseline total CDAI score of ≥220 to ≤250 was considered an IBD responder if a CDAI score of <150 was attained at specified time.
  IBD nonresponder: For UC or CD, a participant who did not fulfil the definition of IBD responder at specified time.
  pMCS score: Sum of 3 subscores (rectal bleeding, stool frequency, and physician's global assessment) excluding endoscopic subscore; ranging from 0 (none) to 9 (severe disease).
  CDAI score: A weighted sum of 8 disease activity variables with scores ranging from 0 to over 600, where higher score = higher disease activity.
  The normal range for sperm concentration is ≥15 million sperm cells/mL.
Time Frame: Baseline to Week 26
Population: Participants in the Week 26 Semen Analysis Set (included all participants who took ≥ 1 dose of study drug and had 2 evaluable samples at baseline and at ≥ 1 postbaseline measurement at/after Week 26 or OL Week 13) with available data were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Filgotinib/DB Filgotinib (Responder): Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase (Part A). At Week 13, participants who were IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B).
- Filgotinib/OL Filgotinib (Nonresponder): Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase (Part A). Participants who were IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib 200 mg, tablet, orally, once daily for up to Week 13 during the OL phase.
- Placebo/DB Placebo (Responder): Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase (Part A). At Week 13, participants who were IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B).
- Placebo/OL Filgotinib (Nonresponder): Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase (Part A). Participants who were IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet a prespecified decrease threshold, entered the OL Phase and received OL filgotinib 200 mg, tablet, orally, once daily for up to Week 13 during the OL phase.
Arm/Group | Filgotinib/DB Filgotinib (Responder) | Filgotinib/OL Filgotinib (Nonresponder) | Placebo/DB Placebo (Responder) | Placebo/OL Filgotinib (Nonresponder)
Number analyzed (Participants) | 40 | 21 | 38 | 17
percentage of participants | 5.0 | 0 | 7.9 | 11.8

3. Secondary Outcome: Change From Baseline in Sperm Total Motility at Week 13
Description: The normal range for sperm total motility is ≥40%.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of motile sperms
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 66 | 67
percentage of motile sperms | -0.3 [-1.6 to 1.7] | 0.4 [-1.3 to 1.5]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Other; Median Difference (Final Values) = -0.2, 95% CI 2-sided [-2.1 to 1.8] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

4. Secondary Outcome: Change From Baseline in Sperm Total Motility at Week 26
Description: IBD responder: For UC, a participant who had a reduction of ≥ 2 in pMCS compared with baseline at specified time. For CD, a participant who had a reduction of ≥ 100 points in total CDAI score compared with baseline at specified time. A participant with a baseline total CDAI score of ≥ 220 to ≤ 250 was considered an IBD responder if a CDAI score of <150 was attained at specified time.
  IBD nonresponder: For UC or CD, a participant who did not fulfil the definition of IBD responder at specified time.
  pMCS score: Sum of 3 subscores (rectal bleeding, stool frequency, and physician's global assessment) excluding endoscopic subscore; ranging from 0 (none) to 9 (severe disease).
  CDAI score: A weighted sum of 8 disease activity variables with scores ranging from 0 to over 600, where higher score = higher disease activity.
  The normal range for sperm total motility is ≥40%.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of motile sperms
Arm/Group | Filgotinib/DB Filgotinib (Responder) | Filgotinib/OL Filgotinib (Nonresponder) | Placebo/DB Placebo (Responder) | Placebo/OL Filgotinib (Nonresponder)
Number analyzed (Participants) | 40 | 21 | 36 | 17
percentage of motile sperms | -2.3 [-4.7 to -0.3] | -1.5 [-5.8 to 2.6] | 0.0 [-3.4 to 2.4] | 0.8 [-7.3 to 5.8]

5. Secondary Outcome: Change From Baseline in Total Sperm Count at Week 13
Description: The normal range for total sperm count is ≥ 39 million sperm cells/ejaculate.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperm cells/ejaculate
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 66 | 67
million sperm cells/ejaculate | -11.6 [-19.8 to 9.7] | -9.5 [-23.8 to 0.6]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Other; Median Difference (Final Values) = 5.7, 95% CI 2-sided [-13.4 to 24.7] — Difference in medians and 95% CI for change from baseline at Week 13 was based on quantile regression

6. Secondary Outcome: Change From Baseline in Total Sperm Count at Week 26
Description: IBD responder: For UC, a participant who had a reduction of ≥ 2 in pMCS compared with baseline at specified time. For CD, a participant who had a reduction of ≥ 100 points in total CDAI score compared with baseline at specified time. A participant with a baseline total CDAI score of ≥ 220 to ≤ 250 was considered an IBD responder if a CDAI score of <150 was attained at specified time.
  IBD nonresponder: For UC or CD, a participant who did not fulfil the definition of IBD responder at specified time.
  pMCS score: Sum of 3 subscores (rectal bleeding, stool frequency, and physician's global assessment) excluding endoscopic subscore; ranging from 0 (none) to 9 (severe disease).
  CDAI score: A weighted sum of 8 disease activity variables with scores ranging from 0 to over 600, where higher score = higher disease activity.
  The normal range for total sperm count is ≥ 39 million sperm cells/ejaculate.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperm cells/ejaculate
Arm/Group | Filgotinib/DB Filgotinib (Responder) | Filgotinib/OL Filgotinib (Nonresponder) | Placebo/DB Placebo (Responder) | Placebo/OL Filgotinib (Nonresponder)
Number analyzed (Participants) | 40 | 21 | 38 | 17
million sperm cells/ejaculate | 2.0 [-19.6 to 17.2] | -4.6 [-42.3 to 18.3] | -4.1 [-39.8 to 15.9] | 12.7 [-61.4 to 40.8]

7. Secondary Outcome: Change From Baseline in Sperm Concentration at Week 13
Description: The normal range for sperm concentration is ≥15 million sperm cells/mL.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperm cells/mL
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 66 | 67
million sperm cells/mL | 1.0 [-2.2 to 3.9] | 0.7 [-2.7 to 1.7]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Other; Median Difference (Final Values) = 1.0, 95% CI 2-sided [-2.8 to 4.9] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

8. Secondary Outcome: Change From Baseline in Sperm Concentration at Week 26
Description: IBD responder: For UC, a participant who had a reduction of ≥ 2 in pMCS compared with baseline at specified time. For CD, a participant who had a reduction of ≥ 100 points in total CDAI score compared with baseline at specified time. A participant with a baseline total CDAI score of ≥ 220 to ≤ 250 was considered an IBD responder if a CDAI score of <150 was attained at specified time.
  IBD nonresponder: For UC or CD, a participant who did not fulfil the definition of IBD responder at specified time.
  pMCS score: Sum of 3 subscores (rectal bleeding, stool frequency, and physician's global assessment) excluding endoscopic subscore; ranging from 0 (none) to 9 (severe disease).
  CDAI score: A weighted sum of 8 disease activity variables with scores ranging from 0 to over 600, where higher score = higher disease activity.
  The normal range for sperm concentration is ≥15 million sperm cells/mL.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperm cells/mL
Arm/Group | Filgotinib/DB Filgotinib (Responder) | Filgotinib/OL Filgotinib (Nonresponder) | Placebo/DB Placebo (Responder) | Placebo/OL Filgotinib (Nonresponder)
Number analyzed (Participants) | 40 | 21 | 38 | 17
million sperm cells/mL | 1.2 [-3.2 to 10.8] | -0.6 [-8.5 to 23.0] | 0.8 [-2.4 to 5.3] | -3.7 [-11.1 to 15.7]

9. Secondary Outcome: Change From Baseline in Ejaculate Volume at Week 13
Description: The normal range for ejaculate volume is ≥1.5 mL.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: mL
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 66 | 67
mL | -0.2 [-0.3 to 0.1] | -0.1 [-0.3 to 0.0]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Other; Median Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

10. Secondary Outcome: Change From Baseline in Ejaculate Volume at Week 26
Description: IBD responder: For UC, a participant who had a reduction of ≥ 2 in pMCS compared with baseline at specified time. For CD, a participant who had a reduction of ≥ 100 points in total CDAI score compared with baseline at specified time. A participant with a baseline total CDAI score of ≥ 220 to ≤ 250 was considered an IBD responder if a CDAI score of <150 was attained at specified time.
  IBD nonresponder: For UC or CD, a participant who did not fulfil the definition of IBD responder at specified time.
  pMCS score: Sum of 3 subscores (rectal bleeding, stool frequency, and physician's global assessment) excluding endoscopic subscore; ranging from 0 (none) to 9 (severe disease).
  CDAI score: A weighted sum of 8 disease activity variables with scores ranging from 0 to over 600, where higher score = higher disease activity.
  The normal range for ejaculate volume is ≥1.5 mL.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: mL
Arm/Group | Filgotinib/DB Filgotinib (Responder) | Filgotinib/OL Filgotinib (Nonresponder) | Placebo/DB Placebo (Responder) | Placebo/OL Filgotinib (Nonresponder)
Number analyzed (Participants) | 40 | 21 | 38 | 17
mL | 0.0 [-0.5 to 0.2] | -0.3 [-0.8 to 0.2] | -0.2 [-0.5 to 0.1] | -0.1 [-0.7 to 0.4]

11. Secondary Outcome: Change From Baseline in Percent Normal Sperm Morphology at Week 13
Description: The normal range for percent normal sperm morphology is ≥30% normal sperms.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of normal sperms
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 66 | 67
percentage of normal sperms | 2 [-1 to 4] | 1 [-1 to 2]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Other; Median Difference (Final Values) = 2, 95% CI 2-sided [0 to 4] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

12. Secondary Outcome: Change From Baseline in Percent Normal Sperm Morphology at Week 26
Description: IBD responder: For UC, a participant who had a reduction of ≥ 2 in pMCS compared with baseline at specified time. For CD, a participant who had a reduction of ≥ 100 points in total CDAI score compared with baseline at specified time. A participant with a baseline total CDAI score of ≥ 220 to ≤ 250 was considered an IBD responder if a CDAI score of <150 was attained at specified time.
  IBD nonresponder: For UC or CD, a participant who did not fulfil the definition of IBD responder at specified time.
  pMCS score: Sum of 3 subscores (rectal bleeding, stool frequency, and physician's global assessment) excluding endoscopic subscore; ranging from 0 (none) to 9 (severe disease).
  CDAI score: A weighted sum of 8 disease activity variables with scores ranging from 0 to over 600, where higher score = higher disease activity.
  The normal range for percent normal sperm morphology is ≥30% normal sperms.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of normal sperms
Arm/Group | Filgotinib/DB Filgotinib (Responder) | Filgotinib/OL Filgotinib (Nonresponder) | Placebo/DB Placebo (Responder) | Placebo/OL Filgotinib (Nonresponder)
Number analyzed (Participants) | 40 | 21 | 38 | 17
percentage of normal sperms | 3 [1 to 5] | 1 [-2 to 3] | 2 [-4 to 5] | 2 [-2 to 3]

ADVERSE EVENTS:
Time Frame: From first dose up to Week 226
Description: All on-treatment safety data during the study were reported under the treatment received at the onset of the event (As-treated set).
Groups:
- Filgotinib: Participants received filgotinib 200 mg tablet, orally once daily (OD) up to Week 13 in DB phase (Part A). At Week 13, IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B). IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet prespecified decrease threshold, entered the OL Phase, and received OL filgotinib 200 mg, tablet orally OD for up to Week 13 during the OL phase. At Week 26/OL Week 13, IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet prespecified decrease threshold, continued receiving the same study drug they were responding to, as part of LTE for up to 195 weeks. Participants who met prespecified sperm decrease threshold(s) discontinued study drug and switched to SOC regimen selected by investigator and entered the MP for up to 52 weeks.
- Placebo: Participants received placebo (matched to filgotinib) tablet, orally OD up to Week 13 in DB phase (Part A). At Week 13, IBD responders, without meeting pre-specified sperm decrease thresholds, continued DB phase treatment up to Week 26 (Part B). IBD non-responders at Week 13 (end of Part A) or had disease worsening after Week 13 and prior to Week 26 (in Part B), and whose sperm parameters did not meet prespecified decrease threshold, entered the OL Phase, and received OL filgotinib 200 mg, tablet orally OD for up to Week 13 during the OL phase. At Week 26/OL Week 13, IBD responders and who had not experienced disease worsening, and whose sperm parameters did not meet prespecified decrease threshold, continued receiving the same study drug they were responding to, as part of LTE for up to 195 weeks. Participants who met prespecified sperm decrease threshold(s) discontinued study drug and switched to SOC regimen selected by investigator and entered the MP for up to 52 weeks.
Arm/Group | Filgotinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/70
Serious Adverse Events (participants affected / at risk) | 3/92 | 2/70
Other Adverse Events (participants affected / at risk) | 47/92 | 24/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib (N=92) | Placebo (N=70)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib (N=92) | Placebo (N=70)
Colitis ulcerative (Gastrointestinal disorders) | 14 | 3
Latent tuberculosis (Infections and infestations) | 5 | 5
Nasopharyngitis (Infections and infestations) | 17 | 3
COVID-19 (Infections and infestations) | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Furuncle (Infections and infestations) | 1 | 4
Headache (Nervous system disorders) | 7 | 0
Pyrexia (General disorders) | 5 | 4
Gastritis (Gastrointestinal disorders) | 7 | 1

LIMITATIONS AND CAVEATS:
The study was terminated based on the sponsor's decision for reasons other than safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03201445/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT03201445/SAP_001.pdf